CLINICAL TRIAL: NCT00438165
Title: Age 12 Follow-up of Early Preventive Intervention
Brief Title: Age 12 Follow-up of Early Preventive Intervention (Memphis)
Acronym: MemphisY12
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 02-0683; R01MH068790 (NIH)
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Child Rearing; Reproductive Behavior; Risk Reduction Behavior
Keywords: nurse; home visits; pregnancy; welfare; child development
MeSH Terms: conditions — Reproductive Behavior; Risk Reduction Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): Control group
- 2 (Experimental): Nurse home visits
  Interventions: Behavioral: home visitation

INTERVENTIONS:
Behavioral: home visitation — Home visitation by nurses from midway through pregnancy until child age 12
  Arms: 2

SUMMARY:
To examine the impact of prenatal and infancy home visiting by nurses from child age 2 through 12.

DETAILED DESCRIPTION:
This study is a longitudinal follow-up of 679 low-income women (89% African American) and their firstborn and subsequent children who have participated in a randomized trial of prenatal and infancy home visiting by nurses in Memphis, Tennessee since 1988. The study was conducted when the first-born children completed sixth grade, at around their 12th birthday.

The current follow-up was designed to determine whether: a) nurse-visited women differ from comparison group women in their life-course outcomes (the number and spacing of subsequent pregnancies and births; the rates of marriage and cohabitation with the father of the child; their employment, career growth, economic self-sufficiency, and welfare dependence; and behavioral problems due to substance abuse; arrests for serious misdemeanors and felonies); b) children of nurse-visited women differ from comparison-children in their academic achievement, placements in special education, rates of grade retention, conduct in school, and academic achievement; c) there are lower rates of developmental disability, grade retention, placement in special education, and school disciplinary actions among subsequent children born to nurse-visited women; d) nurse-visited families have fewer government expenditures and higher taxes paid; e) the effects of the program on child outcomes are concentrated on children born to women with low psychological resources; f) the effects of the program on maternal life course and government costs are concentrated on women with high psychological resources; g) the effects of the program on children are greater in schools and neighborhoods that contain greater risks for academic and behavioral problems; h) the effect of the program on children's disruptive behavior problems is explained by the combined effects of the program on maternal life-course, qualities of parental care-giving, and children's sequential processing skills, and aggressive and violent themes, reliance on adults, and story incoherence in their responses to the McArthur Story Stem Battery at earlier assessments. Data will be derived from maternal interviews and reviews of state administrative and school records. Results from this trial will provide policy makers with an estimate of likely long-term effects of this program when it is conducted in close to real-life conditions.

ELIGIBILITY:
Inclusion Criteria:

* Women <29 weeks gestation
* No previous live births
* At least 2 socio-demographic risk characteristics; e.g. unmarried, <12 years of education, unemployed.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 609 (Actual)
Dates: Start 2003-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
the number and spacing of subsequent pregnancies and births | When first child is 12
the rates of marriage and cohabitation with the father of the child | When first child is 12
mothers' employment, career growth, economic self-sufficiency, and welfare dependence | When first child is 12
mothers' behavioral problems due to substance abuse | When first child is 12
children's academic achievement, placements in special education, rates of grade retention, conduct in school, and academic achievement | At age 12
rates of developmental disability, grade retention, placement in special education, and school disciplinary actions among subsequent children | At age 12
mothers' arrests for serious misdemeanors and felonies | When first child is 12

CONTACTS AND LOCATIONS:
Overall Officials: David L Olds, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Rochester School of Nursing, Rochester, New York, United States

REFERENCES:
- [Background] Olds DL, Kitzman H, Cole R, Robinson J, Sidora K, Luckey DW, Henderson CR Jr, Hanks C, Bondy J, Holmberg J. Effects of nurse home-visiting on maternal life course and child development: age 6 follow-up results of a randomized trial. Pediatrics. 2004 Dec;114(6):1550-9. doi: 10.1542/peds.2004-0962. PMID 15574614
- [Background] Kitzman H, Olds DL, Sidora K, Henderson CR Jr, Hanks C, Cole R, Luckey DW, Bondy J, Cole K, Glazner J. Enduring effects of nurse home visitation on maternal life course: a 3-year follow-up of a randomized trial. JAMA. 2000 Apr 19;283(15):1983-9. doi: 10.1001/jama.283.15.1983. PMID 10789666
- [Background] Kitzman H, Olds DL, Henderson CR Jr, Hanks C, Cole R, Tatelbaum R, McConnochie KM, Sidora K, Luckey DW, Shaver D, Engelhardt K, James D, Barnard K. Effect of prenatal and infancy home visitation by nurses on pregnancy outcomes, childhood injuries, and repeated childbearing. A randomized controlled trial. JAMA. 1997 Aug 27;278(8):644-52. PMID 9272896
- [Background] Olds DL, Kitzman H, Hanks C, Cole R, Anson E, Sidora-Arcoleo K, Luckey DW, Henderson CR Jr, Holmberg J, Tutt RA, Stevenson AJ, Bondy J. Effects of nurse home visiting on maternal and child functioning: age-9 follow-up of a randomized trial. Pediatrics. 2007 Oct;120(4):e832-45. doi: 10.1542/peds.2006-2111. PMID 17908740
- [Derived] Olds DL, Kitzman HJ, Cole RE, Hanks CA, Arcoleo KJ, Anson EA, Luckey DW, Knudtson MD, Henderson CR Jr, Bondy J, Stevenson AJ. Enduring effects of prenatal and infancy home visiting by nurses on maternal life course and government spending: follow-up of a randomized trial among children at age 12 years. Arch Pediatr Adolesc Med. 2010 May;164(5):419-24. doi: 10.1001/archpediatrics.2010.49. PMID 20439792
- [Derived] Kitzman HJ, Olds DL, Cole RE, Hanks CA, Anson EA, Arcoleo KJ, Luckey DW, Knudtson MD, Henderson CR Jr, Holmberg JR. Enduring effects of prenatal and infancy home visiting by nurses on children: follow-up of a randomized trial among children at age 12 years. Arch Pediatr Adolesc Med. 2010 May;164(5):412-8. doi: 10.1001/archpediatrics.2010.76. PMID 20439791